CLINICAL TRIAL: NCT05587075
Title: Clinical Effect and Safety Analysis of Liu Yingmin Long Round Needle in the Treatment of Cervical Spondylotic Radiotelegraphy and Its Effect on Pain and Functional Recovery
Brief Title: Clinical Effect of Long Round Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhanqing Xie (Other)
Responsible Party: Sponsor-Investigator, Zhanqing Xie, Deputy chief physician, The No. 2 Hospital of Baoding
Organization: The No. 2 Hospital of Baoding (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HBaoding
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Cervical Spondylotic Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group was treated with filiform needle.
  Interventions: Procedure: Filiform needle
- Observation group (Experimental): The observation group was treated with long round needle.
  Interventions: Procedure: Long round needle

INTERVENTIONS:
Procedure: Filiform needle — A needle treatment: guide patients take lying or sitting, keep relaxed, select Jingjiaji Point, Fengchi Point, Jianjing Point, Tianzhu Point, Houxi point, Hegu Point, Waiguan Point, preoperative, marker points, conventional disinfection, application specification of 0.35mmx50mm disposable sterile acupuncture needle, in the marker quick needle subcutaneous, slow needle to feel acid swelling feeling, keep needle 30min, once a day, last 5d for 1 course, a total of 4 courses of treatment.
  Arms: Control group
Procedure: Long round needle — Long round needle treatment: mark tendon lesions, take 3-5 tendon lesion points for needle point, after injection of 0.5% lidocaine 1mL, local anesthesia, to hold long round needle, slowly hierarchical detection to tendon lesion points, patients feel acid, hemp, swelling feeling is appropriate, to close method line knot treatment: straight to tendon lesions point surface, scraping, to remove the surface adhesion. Do not cross the superficial surface of the clavicle, sternocleidomastoid muscle deep surface, gentle action. After the needle was released, the pinhole was covered with a disposable dressing, bandaged for 2d, once a week, once for 1 course, and for a total of 4 courses of treatment.
  Arms: Observation group

SUMMARY:
The goal of this clinical trial is to test in the clinical effect of long round needle in the treatment of cervical spondylotic radiculopathy, and analyze its safety and its influence on pain and functional recovery. The main question it aims to answer is whether long round needle therapy for patients with cervical spondylotic radiculopathy is effective and safe. Participants will be selected as the research objects. They will randomly divided into control group (n = 49) and observation group (n = 49). The control group was treated with filiform needle, and the observation group was treated with long round needle. Researchers will compare the two groups to see the differences on the therapeutic effect, safety, Neck dysfunction index (NDI), pain score (McGill pain questionnaire, MPQ), quality of life (Generic Quality of Life Inventory-74, GQOL-74), and levels of inflammatory factors.

ELIGIBILITY:
Inclusion Criteria:

(1) meet the efficacy criteria for disease certificate diagnosis of Traditional Chinese medicine[4]In the category of "Arthralgia Syndrome" and "Stiff neck", the main diseases: numbness and pain in the shoulder, neck and upper limbs, secondary diseases: unfavorable neck movement, hard, heavy head, thin coating, reddish tongue; (2) cervical X-ray shows hyperplasia of the vertebral body; (3) the patient or family members are informed and signed consent.

Exclusion Criteria:

(1) patients with severe periarthritis of shoulder and mixed cervical spondylosis; (2) spinal canal space-occupying lesions and cervical spine tumors; (3) serious immune system diseases and infectious diseases; (4) liver and kidney insufficiency; (5) cardiovascular and cerebrovascular diseases; (6) mental diseases or medical history; (6) patients with incomplete clinical data and poor compliance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Neck dysfunction index (NDI) | Before treament
  Neck dysfunction index (NDI) was used, with 10 items, 0-5 points for each item, and the total score was 0-50 points. The score value was inversely related to the patient's cervical spine function.
Neck dysfunction index (NDI) | Through study completion, an average of 1 year and 10 months
  Neck dysfunction index (NDI) was used, with 10 items, 0-5 points for each item, and the total score was 0-50 points. The score value was inversely related to the patient's cervical spine function.
McGill pain questionnaire (MPQ) score | Before treament
  Neck dysfunction index (NDI) was used, with 10 items, 0-5 points for each item, and the total score was 0-50 points. The score value was inversely related to the patient's cervical spine function.
McGill pain questionnaire (MPQ) score | Through study completion, an average of 1 year and 10 months
  Neck dysfunction index (NDI) was used, with 10 items, 0-5 points for each item, and the total score was 0-50 points. The score value was inversely related to the patient's cervical spine function.
comprehensive assessment questionnaire (GQOL-74) scale | Before treament
  Using the comprehensive assessment questionnaire (GQOL-74) scale, mainly including psychological function, social function, physical function and other items, the score value is positively correlated with the quality of life of patients.
comprehensive assessment questionnaire (GQOL-74) scale | Through study completion, an average of 1 year and 10 months
  Using the comprehensive assessment questionnaire (GQOL-74) scale, mainly including psychological function, social function, physical function and other items, the score value is positively correlated with the quality of life of patients.
interleukin-8 (IL-8) level | Before treament
  5mL of fasting venous blood was extracted from the two groups before and after treatment, centrifuged at 3000 r/min and 8cm for 10 min.
interleukin-8 (IL-8) level | Through study completion, an average of 1 year and 10 months
  5mL of fasting venous blood was extracted from the two groups before and after treatment, centrifuged at 3000 r/min and 8cm for 10 min.
interleukin-10 (IL-10) level | Before treament
  5mL of fasting venous blood was extracted from the two groups before and after treatment, centrifuged at 3000 r/min and 8cm for 10 min.
interleukin-10 (IL-10) level | Through study completion, an average of 1 year and 10 months
  5mL of fasting venous blood was extracted from the two groups before and after treatment, centrifuged at 3000 r/min and 8cm for 10 min.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhanqing, Baoding, Hebei, China